CLINICAL TRIAL: NCT03637231
Title: Ultra-low-dose Coronary Artery Calcium Scoring: Evaluation of Prognostic Performance and Impact of Physiological Factors on Quantification in a Large Population
Brief Title: Ultra-low-dose CACS in a Large Population
Acronym: ULDCACSLARGE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The preliminary findings render it very unlikely that the methodology can be refined further in order to yield more accurate results even if more patients would be included and the study would be continued.
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: USZ-2017-01158
Record Dates: First submitted 2018-07-26; First posted 2018-08-17 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Standard and ultra-low-dose CAC scoring (Other)
  Interventions: Diagnostic Test: Ultra low-dose CTAC

INTERVENTIONS:
Diagnostic Test: Ultra low-dose CTAC — All patients undergo two non-contrast enhanced CT scans with standard dose (i.e. 120 kVp), one with 80 kVp and one with 70 kVp.

SUMMARY:
Radiation exposure to patients from CT for CAC scoring has steadily decreased in recent years. This is mainly achieved through lowering tube currents alongside with the introduction of iterative reconstruction algorithms which allow compensating for increased image noise. However, the greatest radiation dose reduction can be obtained by reducing peak tube voltage. Yet lowering peak tube voltage remains challenging because tissue attenuation is closely related to photon energy, thus rendering the established thresholds for calculating CAC scores (i.e. Agatston scores) incomparable if peak tube voltages other than the standard 120 kilovolt peak (kVp) are applied. The investigators have developed novel tube-adapted thresholds for CAC scoring by CT at 80 kVp and 70-kVp tube voltage and have shown that these novel thresholds are valid, yielding results closely comparable to the standard 120-kVp protocol. The present study aims to optimize application of such low-dose scans in a general population through assessment of the impact of physiological patient parameters on image parameters such as image noise which per se may impact the accuracy and feasibility of ultra-low-dose CAC scoring with reduced tube voltage. Furthermore, the prognostic performance of such low-dose CAC scoring will be elucidated.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for a non-contrast enhanced CT scan for CAC scoring
* Male and Female subjects ≥18 years of age,
* Written informed consent

Exclusion Criteria:

* Pregnancy or breast-feeding
* CACS of 0 after inclusion of 50 patients with CACS 0 (as assessed visually after the first CT scan, prior to performing the 3 additional study scans)
* History of coronary artery stenting, coronary artery bypass grafting, of implantation of cardiac devices (e.g. valve prosthesis, pacemaker, implantable cardioverter defibrillator etc.)
* Enrolment of the investigator, his/her family members, employees and other dependent persons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2018-07-05 (Actual); Primary Completion 2021-10-25 (Actual); Study Completion 2021-10-25 (Actual)

PRIMARY OUTCOMES:
Impact of BMI on CAC scores derived from low-dose versus standard-dose CT | 2 years
  Assessment of deviation of CAC scores derived from low-dose CT versus standard-dose CT (i.e. standard of reference) by calculating bias and Bland-Altmann limits of agreement as well as intraclass correlation in different subgroups of patients, stratified by body mass index.

SECONDARY OUTCOMES:
Prognostic value of CAC scores derived from CT scans with varying tube voltages | 2 years
  Assessment of sensitivity and specificity CAC scores derived from low-dose CT versus standard-dose CT (i.e. standard of reference) to predict future cardiovascular events (i.e. myocardial infarction, revascularisation, death) over a short to mid-term follow-up period (i.e. 2 years).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nuclear Medicine, University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grani C, Vontobel J, Benz DC, Bacanovic S, Giannopoulos AA, Messerli M, Grossmann M, Gebhard C, Pazhenkottil AP, Gaemperli O, Kaufmann PA, Buechel RR. Ultra-low-dose coronary artery calcium scoring using novel scoring thresholds for low tube voltage protocols-a pilot study. Eur Heart J Cardiovasc Imaging. 2018 Dec 1;19(12):1362-1371. doi: 10.1093/ehjci/jey019. PMID 29432592
- [Derived] Bechtiger FA, Grossmann M, Bakula A, Patriki D, von Felten E, Fuchs TA, Gebhard C, Pazhenkottil AP, Kaufmann PA, Buechel RR. Risk stratification using coronary artery calcium scoring based on low tube voltage computed tomography. Int J Cardiovasc Imaging. 2022 Oct;38(10):2227-2234. doi: 10.1007/s10554-022-02615-x. Epub 2022 Apr 23. PMID 37726457
- [Derived] Sartoretti T, Gennari AG, Sartoretti E, Skawran S, Maurer A, Buechel RR, Messerli M. Fully automated deep learning powered calcium scoring in patients undergoing myocardial perfusion imaging. J Nucl Cardiol. 2023 Feb;30(1):313-320. doi: 10.1007/s12350-022-02940-7. Epub 2022 Mar 17. PMID 35301677